CLINICAL TRIAL: NCT04827147
Title: Randomized Controlled Multicenter Clinical Trial of Multi-Periscopic Prism Glasses for Homonymous Hemianopia
Brief Title: Clinical Trial of Multi-Periscopic Prism Glasses for Hemianopia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Eli Peli, Senior Scientist, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MPPvsFPP; R01EY023385 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Homonymous Hemianopia
MeSH Terms: conditions — Hemianopsia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MPP first, FPP second (Experimental): Participants in this arm will receive the MPP in the first period of the crossover and the FPP in the second period.
  Interventions: Device: Multi-Periscopic Prism (MPP) glasses; Device: Fresnel Peripheral Prism (FPP) glasses
- FPP first, MPP second (Experimental): Participants in this arm will receive the FPP in the first period of the crossover and the MPP in the second period.
  Interventions: Device: Multi-Periscopic Prism (MPP) glasses; Device: Fresnel Peripheral Prism (FPP) glasses

INTERVENTIONS:
Device: Multi-Periscopic Prism (MPP) glasses — Spectacles with multi-periscopic prisms mounted as oblique peripheral prism segments
Device: Fresnel Peripheral Prism (FPP) glasses — Spectacles with conventional permanent Fresnel prisms mounted as oblique peripheral prism segments

SUMMARY:
This clinical trial will evaluate the efficacy of two types of high-power prism glasses that provide field of view expansion for patients with homonymous hemianopia (the complete loss of half the field of vision on the same side in both eyes).

DETAILED DESCRIPTION:
Patients with hemianopic field loss may be unaware of objects in their blind (non-seeing) hemi-field and often experience difficulties with hazards, such as walking into obstacles on the side of the field loss. Prism glasses that provide field of view expansion may be helpful in detecting hazards on the blind side. In this clinical trial, two types of high power prism glasses will be evaluated. A new design of prisms, Multi-Periscopic Prisms (MPP), will be compared to commercially-available permanent Fresnel peripheral prism (FPP) glasses. The extent to which the prismatic devices improve detection of hazards on the side of the field loss and are helpful when walking will be evaluated.

Participants will try each type of prism glasses at home for 4 weeks in counterbalanced order. Prism glasses will be fitted by Low Vision Practitioners at vision rehabilitation clinics. Participants will attend in-office study visits before and after wearing each type of prism glasses. At the in-office visits they will complete a test that involves detecting pedestrian hazards in a video simulating a walk through a busy shopping mall (virtual reality, VR, walking simulator test). In addition, they may be asked to complete questionnaires to record their experiences of using the prism glasses.

After wearing the second pair of prism glasses, participants will be asked to complete a questionnaire comparing the two types of prism glasses and to select their preferred type. A clinical decision will be made as to whether the participant should continue to use either the first or second pair of prism glasses (e.g. if a participant finds one pair of prism glasses helpful for obstacle avoidance when walking). For participants who continue with the prism glasses, telephone follow-up interviews will be conducted after about 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Homonymous hemianopia with or without macular sparing for at least 3 months
* Visual acuity of at least 20/50 in each eye, with correction if needed
* Refractive error in the -12D to +5D range
* Able to walk independently, using a cane or walker if needed
* Able to communicate in English sufficiently to understand the study procedures and how to use the prisms

Exclusion Criteria:

* Central visual field loss in the seeing hemifield of either eye (e.g. from macular degeneration, glaucoma, diabetic retinopathy or other maculopathies)
* Hemi-spatial neglect
* Significant cognitive impairment
* Dementia
* Any other physical or mental disabilities, or general health problems that could impair the ability to be independently mobile (i.e., walk ), participate in the VR walking simulator test or use the prism glasses

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in blind-side detection rate for hazards approaching at a bearing angle of 40 degrees | After 4 weeks of wearing first pair of prism glasses, After 4 weeks of wearing second pair of prism glasses
  Improvement in detection rate with prism glasses for hazards approaching from the blind side at a bearing angle of 40 degrees in the VR walking simulator test. Improvement is a binary outcome, defined as blind-side detection rate (number of pedestrians detected as a percentage of the total number of pedestrian events) which is significantly higher (z-test for two proportions) with than without prism glasses at the same visit.

SECONDARY OUTCOMES:
Device preference | After 4 weeks of wearing the second pair of prism glasses
  Number of participants selecting each device as a percentage of the total number of participants enrolled
Improvement in blind-side detection rate for hazards approaching at a bearing angle of 20 degrees | After 4 weeks of wearing first pair of prism glasses, After 4 weeks of wearing second pair of prism glasses
  Improvement in detection rate with prism glasses for hazards approaching from the blind side at a bearing angle of 20 degrees in the VR walking simulator test. Improvement is a binary outcome, defined as blind-side detection rate (number of pedestrians detected as a percentage of the total number of pedestrian events) which is significantly higher (z-test for two proportions) with than without prism glasses at the same visit.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Peli, OD MSc, Principal Investigator — Schepens Eye Research Institute of Massachusetts Eye and Ear
Locations (8):
- United States (8):
  - UAB Center for Low Vision Rehabilitation, Callahan Eye Hospital, Birmingham, Alabama
  - UCHealth Sue Anschutz-Rodgers Eye Center, Denver, Colorado
  - Visual Health and Surgical Center, Palm Springs, Florida
  - Illinois College of Optometry, Chicago, Illinois
  - Schepens Eye Research Institute, Boston, Massachusetts
  - New England College of Optometry, Boston, Massachusetts
  - The Eye and Vision Center at MCPHS, Worcester, Massachusetts
  - UMass Chan Medical School, Worcester, Massachusetts